CLINICAL TRIAL: NCT03568370
Title: Effects of Olive Oil on Nipple Cracking, Nipple Pain and Maternal Satisfactions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Lin, Chen-xi, PI, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-106-05-131
Record Dates: First submitted 2017-10-11; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cracked Nipple During Lactation
MeSH Terms: interventions — Olive Oil; Milk, Human

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olive oil (Experimental): use one drop olive oil on each nipple after each feeding
  Interventions: Other: olive oil
- breast milk (No Intervention): use breast milk on each nipple after each feeding

INTERVENTIONS:
Other: olive oil — Evaluate the effectiveness of olive oil and human milk in the prevention of nipple cracking, nipple pain and maternal satisfaction in lactating women during the first 3 days of treatment and the 7th and 10th day after delivery.
  Other Names: human milk
  Arms: olive oil

SUMMARY:
The aim of the study is to evaluate the effectiveness of olive oil in the prevention of nipple cracking, nipple pain and ascension maternal satisfaction in lactating women. It's a prospective, randomized study of 80 lactating women, admitted to Tri-Service General hospital postpartum unit. Eligible patients were randomized to olive oil group or breast milk group and evaluate the effect of olive oil for nipple pain, nipple trauma, and maternal satisfaction.

DETAILED DESCRIPTION:
Previous studies have shown that olive oil, applied to the skin, has analgesic and anti-inflammatory properties. It is proposed in this study that olive oil may also help prevent cracked nipple and sore nipple in breastfeeding mothers. The aim of the study is to evaluate the effectiveness of olive oil in the prevention of nipple cracking, nipple pain and ascension of maternal satisfaction in lactating women. It's a prospective, randomized study of 80 lactating women, admitted to TSGH postpartum unit. Eligible patients were randomized into two groups of 40 women. In Group 1 Olive oil will be applied on the nipple after breastfeeding, and in Group 2 drops of breast milk were applied to the nipple after feeding. Clinical evaluations were made during the first 3 days of treatment and the 7th and 10th day after delivery. Furthermore, we will check the 1month breastfeeding rate data, which collected by the hospital nurse for baby-friendly hospital policy.

ELIGIBILITY:
Inclusion Criteria:

* Normal spontaneous delivery.
* Pregnancy weeks between 37-42.
* Single birth.
* Initiated breastfeeding.

Exclusion Criteria:

* Presence of crack in the nipple.
* Medication applied to the nipple
* The maternal health condition that may interfere with breastfeeding.
* The infant with congenital abnormalities that would impair breastfeeding.
* The infant attained low birth weight or other criteria to intensive care unit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Nipple pain change | Change from baseline nipple pain at 10 days
  use Numeric Rating Scale 0-10 point
Nipple sore change | Change from baseline nipple pain at 10 days
  use Nipple Soreness Score 0-5 point
Nipple trauma change | Change from baseline nipple trauma at 10 days
  use Nipple Trauma Score 0-5 point
breastfeeding duration | 30 days
  use Infant Feeding Categories

SECONDARY OUTCOMES:
Maternal satisfaction | baseline from Baseline nipple sore at 10 days
  use Maternal Satisfaction Questionnaire 0-40 point

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Xi Lin, Study Chair — lin050027@hotmail.com
Locations (1):
- Lin, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin CX, Lu YY. Comparative Effectiveness of Olive Oil and Breast Milk on Nipple Soreness in Breastfeeding Mothers. Breastfeed Med. 2023 Oct;18(10):779-784. doi: 10.1089/bfm.2023.0081. Epub 2023 Oct 5. PMID 37797219